CLINICAL TRIAL: NCT06587022
Title: Delineation of Target Volume of Stereotactic Radiotherapy for Spinal Tumors
Acronym: ST-SBRT
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ST-SBRT
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Spinal Tumor
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group 1: Group 1(small target delineation)：The target bolume only includes local tumor.
  Interventions: Radiation: Target volume delineation
- group 2: Group 2(small target delineation)：The target bolume includes local tumor and adjacent vertebral area.
  Interventions: Radiation: Target volume delineation

INTERVENTIONS:
Radiation: Target volume delineation — Group 1(small target delineation)：The target bolume only includes local tumor. Group 2(small target delineation)：The target bolume includes local tumor and adjacent vertebral area.

SUMMARY:
The purpose of this study was to compare efficacy and side effects of two target delineation methods for stereotactic radiotherapy of metastatic spinal tumors.

DETAILED DESCRIPTION:
The purpose of this study was to compare efficacy and side effects of two target delineation methods for stereotactic radiotherapy of metastatic spinal tumors. This is a bidirectional cohort study planned to enroll approximately 500 patients with metastatic spinal tumors. Patients are divided into two groups according to the target delineation method. Group 1：The target bolume only includes local tumor. Group 2：The target bolume includes local tumor and adjacent vertebral area.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spinal metastases or primary tumors receiving stereotactic radiotherapy;
* Patients with sufficent pre-treatment imaging data
* Patients who can cooperate with imaging review and follow-up after radiotherapy.

Exclusion Criteria:

* Patients with an expected survival of less than 3 months;
* Patients with second-course radiotherapy;
* Patients with physical conditions that cannot tolerate stereotactic radiotherapy;
* Patients with extensive spinal metastasis and no local therapeutic value

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant tumor spinal metastasis who received or will receive stereotactic radiotherapy, without preoperation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate（DCR） | 2 years
  Disease Control Rate（DCR），including complete response（CR），partial response(PR) and stable disease(SD ).
Pain relief rate | 3 months
  VAS Score(Visual Analog Scale Score) decreased after treatment

SECONDARY OUTCOMES:
Incidence of side effects | 2 years
  radiation myelitis,radiation esophagitis, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqing Zhuang, Study Director — Peking University Third Hospital
Locations (1):
- Department of Radiation Oncology Cancer Center, Peking University Third Hospital 49# North Garden Rd.,Haidian Dist., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No